CLINICAL TRIAL: NCT02038465
Title: REMEDIATION COGNITIVE DE LA MÉMOIRE AUTOBIOGRAPHIQUE DANS LA SCHIZOPHRENIE AU MOYEN DE SENSECAM
Brief Title: Cognitive Remediation of Autobiographical Memory in Schizophrenia Using SenseCam®
Acronym: RéMABSchiz
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5539
Record Dates: First submitted 2013-06-25; First posted 2014-01-16 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia Cognition Autobiographical Memory Cognitive Remediation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient (Other): Complete questionary remembering the day
  Interventions: Device: Questionary
- healthy volunteers (Other): - Complete questionary, remembering the day
  Interventions: Device: Questionary

INTERVENTIONS:
Device: Questionary — Test the effectiveness of two techniques of cognitive remediation of autobiographical memory using an innovative tool called SenseCam ® for patient
Device: Questionary — Test the effectiveness of two techniques of cognitive remediation of autobiographical memory using an innovative tool called SenseCam ® for healthy volunteers

SUMMARY:
The aim of the study is to assess the efficiency of SenseCam® in patients with schizophrenia by comparing two cognitive remediation methods of autobiographical memory.Patients and control participants will be invited to carry SenseCam® during 7 hours per day minimum and for 4 successive days. Each ending day when carry SenseCam®, they will be asked to go to the laboratory where 4 types of interventions will be successively done according to the randomization: 1) a simple visual retrospective procedure (SVR), 2) a visual retrospective procedure coupled with a specific cueing intervention (VR-SC), 3) a verbal retrospective (VbR) and 4) no intervention (control condition).The testing phase will take place 14 days after the last day of data collection and will consist in a cued recall task and a recognition task using the pictures obtained by the SenseCam® of the participants.According to our hypotheses, the vividness of memories will be higher in events subjected to the VR-SC procedure than in events subjected to the SVR and VbR procedures. This effect is expected for both patients with schizophrenia and controls participants. Since strategies to enrich memory details will be explicitly given to the patients when using the VR-SC procedure, we assume that patients will be able to normalize their scores.

ELIGIBILITY:
Inclusion Criteria:

* for both patients and controls
* male or female willing to participate and who have signed up the legal document
* under the protection of health insurancefor patients only
* schizophrenia or schizo-affective disorder according to the DSM-IV
* TR criteria
* clinically stable for at least 2 monthsfor controls only
* no psychiatric history

Exclusion Criteria:

* for both patients and controls
* current severe or unstable somatic illness
* neurological history (epilepsia, brain injury, brain surgery…)
* current substance use disorder (DSM-IV-TR)
* current major depressive disorder (DSM-IV-TR)
* mental retardation (IQ < 70)
* pregnancy, breast feeding
* current legal controlfor patients only
* treatment comprising benzodiazepines
* benzodiazepines intake during the last 3 weeksfor controls only
* psychotropic intake during the last 3 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Specificity of memories recovered by using the SenseCam camera during the trial | 1 month
  Test the effectiveness of two techniques of cognitive remediation of autobiographical memory using an innovative tool called SenseCam.This specificity will be evaluated by the experimenter by scoring wealth in detail memories reported during the cued recall task

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Berna, MD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Berna, Strasbourg, France